CLINICAL TRIAL: NCT04854759
Title: The Use of Amantadine in the Prevention of Progression and Treatment of COVID-19 Symptoms in Patients Infected With the SARS-CoV-2 Virus
Brief Title: The Use of Amantadine in the Prevention of Progression and Treatment of COVID-19 Symptoms
Acronym: COV-PREVENT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Independent Public Clinical Hospital No. 4 in Lublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUB-COV-2021-01
Record Dates: First submitted 2021-04-17; First posted 2021-04-22 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental)
  Interventions: Drug: Amantadine Hydrochloride
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amantadine Hydrochloride — 100 mg, capsule
  Arms: Study group
Drug: Placebo — 100 mg, capsule
  Arms: Control group

SUMMARY:
The use of amantadine in the prevention of progression and treatment of COVID-19 symptoms in patients infected with the SARS-CoV-2 virus. Multicenter randomized, double-blind, placebo-controlled, non-commercial clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and over
* Can give informed consent
* Confirmed positive result for SARS-CoV-2 within 72 hours from the date the result was issued (according to the laboratory report)
* Patient presently symptomatic with one or more of the following symptoms: fever, cough, myalgia, mild dyspnoea, chest pain, diarrhea, nausea, vomiting, anosmia, lack of taste, sore throat, nasal congestion
* At initial screening, the subject will report at least one and no more than 3 of the following risk factors for clinical worsening: age ≥40, obesity, hypertension, diabetes, pulmonary disease (e.g., asthma, COPD), and immune disorders (e.g. rheumatoid arthritis, lupus), neurological diseases: e.g. after a distant stroke or trauma to the brain, multiple sclerosis, dementia and other neurodegenerative diseases)
* Patients hospitalized due to meeting the above criteria and requiring observation in a hospital or outpatient setting.

Exclusion Criteria:

* Disease severe enough to meet the study's primary endpoint of clinical worsening (eg, current O2 saturation <92% with patient exposure to room air, current use of supplemental oxygen to maintain O2 saturation ≥ 92%).
* WHO score ≥4 (requires oxygen therapy during hospitalization)
* Concomitant diseases which, in the opinion of the attending physician, prevent the patient from participating in the study, such as: decompensated cirrhosis, active ulcer disease, epilepsy and symptomatic convulsions, untreated angle-closure glaucoma determined on the basis of the patient's interview and / or medical documentation . In addition, immunocompromised patients (solid organ transplant, BMT, AIDS, renal failure (patients with renal impairment may develop drug poisoning) or other diseases not mentioned and other diseases treated with biological, immunological and / or steroids in high doses will not be eligible for the study. doses (> 20 mg prednisone daily).
* Hypersensitivity to any component of the preparation, severe congestive heart failure, cardiomyopathy, myocarditis, II-III degree AV block, bradycardia, clinically significant prolongation of the QT interval, or a family history of congenital long QT syndrome, severe ventricular arrhythmias (including torsade de pointes), concomitant use of drugs that prolong the QT interval, hypokalaemia, hypomagnesaemia,
* Pregnancy, the period of breastfeeding.
* Parallel intake of memantine or other drugs acting on the CNS (neuroleptics, anxiolytics, antiepileptic drugs, antidepressants).
* Other neurological conditions with agitation or confusion, delirium syndromes or psychoses.
* Receipt of a partial or full vaccination schedule against SARS-CoV-2 is also an exclusion criterion from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Development of clinical deterioration | Up to day 15 from randomization
  Defined as dyspnoea - physical examination - doctor's assessment
Clinical deterioration occurs | Up to day 15 from randomization
  Defined as drop in O2 saturation (<92% with patient exposure to room air) and / or additional oxygen demand to maintain O2 saturation ≥92%)
Clinical deterioration occurs | Up to day 15 from randomization
  Defined as achievement of ≥4 points on the WHO [OSCI-WHO] scale (7-point clinical status assessment scale)

SECONDARY OUTCOMES:
General Health Scale (PROMIS® Global Health Scale) | Day 15, 30 complementary visit-optional, 90, 150, 210
  Mean Global Health scores for each arm at day 15, 30 complementary visit-optional, 90, 150, 210. PROMIS® instruments are scored using item-level calibrations. This method of scoring uses "response pattern scoring," which uses responses to each item for each participant.
The neurological assessment | Day 15, 30 complementary visit-optional, 90, 150, 210
  will include the assessment of neurological functions based on:
  1. scales for fatigue,
  2. depression,
  3. disorders of smell and taste,
  4. sleep disorders,
  5. quality of life.
Time to clinical deterioration | Day 15, 30 complementary visit-optional, 90, 150, 210
Survival time | Day 15, 30 complementary visit-optional, 90, 150, 210

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Rejdak, Professor, PhD, MD, Principal Investigator — Independent Public Clinical Hospital No. 4 in Lublin
Locations (8):
- Poland (8):
  - Regionalny Szpital Specjalistyczny im. dr Władysława Biegańskiego Oddział Neurologii i Neuroimmunologii Klinicznej, Grudziądz
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej w Kalwarii Zebrzydowskiej, Kalwaria Zebrzydowska
  - Oddział Obserwacyjno-Zakaźny SPSz Woj. Im. Jana Bożego Lublin, Lublin
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Klinika Chorób Wewnętrznych Nefrologii i Endokrynologii Klinicznego Szpitala Wojewódzkiego nr 2 im. Św. Jadwigi Królowej, Rzeszów
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego Szpital Kliniczny Dzieciątka Jezus, Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnętrznych i Administracji w Warszawie, Warsaw
  - Oddział Kardiologiczny Samodzielny Publiczny Zespół Zakładów Opieki Zdrowotnej w Wyszkowie, Wyszków

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rejdak K, Fiedor P, Bonek R, Goch A, Gala-Bladzinska A, Chelstowski W, Lukasiak J, Kiciak S, Dabrowski P, Dec M, Krol ZJ, Papuc E, Zasybska A, Segiet A, Grieb P. The use of amantadine in the prevention of progression and treatment of COVID-19 symptoms in patients infected with the SARS-CoV-2 virus (COV-PREVENT): Study rationale and design. Contemp Clin Trials. 2022 May;116:106755. doi: 10.1016/j.cct.2022.106755. Epub 2022 Apr 4. PMID 35390511